CLINICAL TRIAL: NCT01812317
Title: Effect of Real-fire Training on Vascular Function
Acronym: FIREPROOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11-SS-0086; PG/11/27/28842 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2013-03-04; First posted 2013-03-18 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Vascular Function; Atherothrombosis
Keywords: firefighters; fire-simulation training; myocardial infarction; endothelial function; thrombosis
MeSH Terms: conditions — Thrombosis; Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real-fire training exercise (Active Comparator): Subjects will undergo a 20 minute standardised training exercise in a fire simulation facility.
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber Study
- Sedentary training session (Sham Comparator): Subjects will undergo a training exercise where they will remain sedentary for 20 mins in an ambient temperature.
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber Study

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography to measure forearm blood flow during intra-arterial infusion of the vasodilators Verapamil (10-100 µg/min), bradykinin (100-1000 pmol/min), sodium nitroprusside (2-8 µg/min) and Acetylcholine (5-20 µg/min).
  Other Names: BK; SNP; ACh; VP
Procedure: Badimon Chamber Study — Ex-vivo assessment of thrombus formation using the Badimon Chamber

SUMMARY:
Fire-fighters are at increased risk of death from heart attacks when compared to other emergency service professionals whose jobs involve similar components such as emergency call-outs and shift work. The unique risk to fire-fighters is likely to reflect a combination of factors including extreme physical exertion, mental stress, heat and pollutant exposure.

In the largest analysis of cause of death amongst on-duty fire-fighters, fire-fighter deaths were classified according to the duty performed during the onset of symptoms or immediately prior to any sudden death. The majority of deaths due to a cardiovascular cause (i.e. heart attack) occurred during fire-suppression whilst this activity represented a relatively small amount of a fire-fighters professional time. Fire simulation training centers offer a unique opportunity to assess the heart, blood and blood vessel response to fire suppression in a controlled environment.

In this study the investigators will assess healthy career fire-fighters on two occasions: following a fire-suppression training exercise in a purpose built real-fire training center, and following a sedentary period as a control. The investigators will take blood samples to measure platelet activity (platelets are the particles in blood that help blood clot) and will examine how blood clots outside of the body. The investigators will then perform studies placing small needles in the arm to assess blood vessel function following fire suppression. By undertaking this comprehensive assessment of blood, blood vessel and heart function we hope to understand the mechanisms whereby the risk of a heart attack is influenced by fire suppression. The investigators hypothesize that following the fire-suppression exercise firefighters blood will clot more readily and their blood vessels will not relax properly which are two of the main processes in the development of a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy firefighters

Exclusion Criteria:

* Current smoker
* History of lung or ischaemic heart disease
* Malignant arrhythmia
* Systolic blood pressure >190mmHg or <100mmHg
* Renal or hepatic dysfunction
* Previous history of blood dyscrasia
* Unable to tolerate the supine position
* Blood donation within the last 3 months
* Recent respiratory tract infection within the past 4 weeks
* Routine medication including aspirin and NSAIDs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by venous occlusion plethysmography in response to infused vasodilators | 3-6 hours post exposure

SECONDARY OUTCOMES:
Ex-vivo thrombus formation using the Badimon chamber | 2 hours post exposure
Plasma t-PA and PAI concentrations following infusion of bradykinin | During forearm study, 3-6 hours post exposure

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD PhD, Study Chair — University of Edinburgh; Nicholas L Mills, MBChB PhD, Study Director — University of Edinburgh; Amanda L Hunter, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh Clinical Research Facility, Edinburgh, United Kingdom

REFERENCES:
- [Result] Hunter AL, Shah AS, Langrish JP, Raftis JB, Lucking AJ, Brittan M, Venkatasubramanian S, Stables CL, Stelzle D, Marshall J, Graveling R, Flapan AD, Newby DE, Mills NL. Fire Simulation and Cardiovascular Health in Firefighters. Circulation. 2017 Apr 4;135(14):1284-1295. doi: 10.1161/CIRCULATIONAHA.116.025711. PMID 28373523